CLINICAL TRIAL: NCT06779799
Title: Characterization of "Bamboo" and Other Vocal Cord Lesions Responsible for Dysphonia in Patients With Systemic Autoimmune Diseases.
Brief Title: Characterization of "Bamboo" and Other Vocal Cord Lesions Responsible for Dysphonia in Patients With Systemic Autoimmune Diseases (BAMBOO)
Acronym: BAMBOO
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC24.0332 - BAMBOO
Record Dates: First submitted 2025-01-07; First posted 2025-01-17 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2024-12

CONDITIONS: Dysphonia; Connective Tissue Disease; Vasculitis
MeSH Terms: conditions — Dysphonia; Connective Tissue Diseases; Vasculitis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this multicenter retrospective observational study is to provide an inventory of the specific and non specific cord vocal lesions that can cause dysphonia in patients with systemic autoimmune diseases. The main question it aims to answer is:

* What are the main cord vocal lesions responsible for dysphonia in patients with a systemic autoimmune disease?
* Is there a diagnosis delay regarding those lesions?
* How are those lesions managed? Participants suffering from dysphonia in a context of a systemic autoimmune disease will be identified, with a review of their medical record.

DETAILED DESCRIPTION:
Patients with a systemic autoimmune disease may face to the occurrence of a dysphonia during the course of their disease. Specific etiologies must be sought for, such as "bamboo nodes", previously reported on small series, especially in patients with systemic erythematosus lupus, but also in other connective tissue disease such as Sharp syndrome, primary Sjögren disease and anti-synthetase syndrome. These nodes are made of fibrosis and immune complexes have been described. The treatment relies on vocal reeducation, oral steroids and sometimes surgery. Other irritative factors must be avoided such as stopping tobacco or treating a gastroesophageal reflux. Increasing the immunosuppressive regimen of the autoimmune disease has also been suggested, but the management is not codified due to the rarity of this condition. Rheumatoid nodules of the vocal cords have also been described in rheumatoid arthritis as well as cricoarytenoid joint arthritis. Granuloma of the vocal cords have also been reported in granulomatosis with polyangiitis. Other non specific etiologies should also be sought for such as mucosal ulcerations, submucous edema or hematoma, or vocal cord palsy.

Owing to the rare series of dysphonia reported in a context of systemic auto-immunity, the aim of this retrospective study is to provide an inventory of the specific and non specific lesions that can cause dysphonia in patients with systemic autoimmune diseases, with the assessment of potential diagnosis delays and therapeutics.

Main objective : To characterize the cord vocal lesions responsible for dysphonia in patients with systemic autoimmune diseases.

Secondary objectives :

* To assess the proportion of "bamboo nodes" compared to non specific lesions in patients with a systemic autoimmune disease suffering from dysphonia.
* To identify potential diagnosis delays.
* To describe the management of these lesions.
* To identify risk factors associated with these lesions.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older
* With a systemic autoimmune disease : rheumatoid arthritis, systemic lupus erythematosus, systemic sclerosis, primary Sjogren disease, sarcoidosis, vasculitis, myositis, Still disease, Sharp syndrome.
* Suffering from dysphonia.
* With a cord vocal/laryngeal lesion highlighted.

Exclusion Criteria:

* Patients under the age of 18 years
* Dysphonia due to a cord vocal palsy related to a neurological condition or malignancy
* History of cervical radiation
* History of oro-tracheal intubation
* Laryngeal cancer
* Participation deny
* Impossibility of consent
* Patients with legal protection

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients aged 18 years or older suffering from dysphonia in a context of a systemic autoimmune disease.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Nature of the cord vocal lesion responsible for dysphonia according to the physician (otorhinolaryngologist, rheumatologist or internist) from medical record | between january 2014 and december 2024
  Diagnosis of the lesion responsible for dysphonia will be determined from medical record : medical report of the otorhinolaryngologist and/or laryngoscopy report if available or anatomopathological report in case of biopsy/surgery of the lesion. If no report from the otorhinolaryngologist is found in the record, then the reported diagnosis from the rheumatologist or the internist will be considered.

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Brest, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning three years and ending fifteen years following the final study report completion
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement